CLINICAL TRIAL: NCT00461370
Title: Phase I, Double-Blind, Placebo-Controlled, Ascending, Single-Dose, Safety, Tolerability and Pharmacokinetic Study of SRX251 Capsules in Healthy Female Volunteers
Brief Title: Safety Study of SRX251 Capsules in Healthy Female Volunteers
Acronym: AVN001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azevan Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVN001
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
Keywords: safety; Phase 1; pharmacokinetics; SRX251; Azevan; safety in healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SRX251

SUMMARY:
The purpose of this study is to determine the safety of SRX251 when given orally. The amount of SRX251 in the blood will also be measured. Healthy women, ages 18-50 years who have been surgically sterilized by tubal ligation, will be enrolled in this study.

DETAILED DESCRIPTION:
Vasopressin appears to be a key mediating factor in menstrual pain. This position stems from findings that the hormone, arginine vasopressin (AVP), causes constriction of uterine blood vessels which in turn produces congestion of the uterus resulting in dysmenorrhea. Prior to menses, blood vessels in the uterine wall become engorged with blood. Elevated concentrations of vasopressin acting through V1a receptors cause constriction of both uterine and vascular smooth muscle, contributing to the discomfort and pain of primary dysmenorrhea. Consequently, blockade of these receptors with a selective V1a receptor antagonist would be expected to provide therapeutic benefits to women with primary dysmenorrhea.

SRX251 is a new chemical entity with potent V1a receptor antagonist properties, and an acceptable safety profile as demonstrated in preclinical studies. This study is intended to evaluate the safety and pharmacokinetic profile of a single oral dose of SRX251 in healthy human female volunteers in preparation for further studies of the safety and pharmacological activity in the amelioration of pain associated with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

1. Females of ≥18 and ≤50 years of age who have a regular menstrual cycle between 24-35 days duration.
2. Have a body mass index (BMI) of ≥18.5 and ≤30.
3. In good health as determined by medical history, a baseline physical examination, vital signs, clinical laboratory tests and electrocardiogram (ECG) measurement.
4. Subject has undergone surgical sterilization by tubal ligation.
5. Subject is willing and able to sign written informed consent prior to receipt of any study medication or beginning study procedures.
6. Subject is willing and able to follow instructions, comply with the protocol requirements and make all required study visits.

Exclusion Criteria:

1. Subject is pregnant or nursing.
2. Subject has undergone surgical sterilization by any method other than tubal ligation (e.g., hysterectomy).
3. Positive results for HIV, hepatitis B surface antigen or hepatitis C antibody tests at screening.
4. Positive urine test for drugs of abuse at screening.
5. Any out-of range laboratory value at screening that has not been reviewed, approved and documented as not clinically significant by the Principal Investigator.
6. Supine blood pressure, after resting for 5-10 minutes, outside a systolic blood pressure range of 90-140 mmHg or a diastolic blood pressure outside a range of 50-90 mmHg on two consecutive measurements taken 5 minutes apart.
7. Supine pulse rate, after resting for 5-10 minutes, greater than 100 bpm or lower than 50 bpm on two consecutive measurements taken 5-10 minutes apart.
8. Has taken any alcohol within 48 hours of ANY study-related activities AND cannot abstain from drinking alcohol during the entire duration of the subject's study participation.
9. Has used any tobacco products in the past 12 months.
10. A history of significant drug allergy or systemic allergic disease (e.g., urticaria, atopic dermatitis).
11. A general medical or psychological condition or behavior, including current substance dependence or abuse that, in the opinion of the investigator, might not permit the subject to complete the study or sign the informed consent.
12. Any clinically significant abnormality on screening 12-lead ECG (e.g., heart block, conduction disorders, ventricular and/or atrial arrhythmias).
13. Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Principal Investigator or the Physician Sub-Investigator, would make the subject unsuitable for the study or put them at additional risk.
14. Routine or PRN consumption of medications or herbal supplements that the subject is unable or unwilling to discontinue during the study. Multivitamins may be consumed during the study.
15. Inability to understand or follow study instructions.
16. Known allergy or hypersensitivity to the investigational study drug/placebo components.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
safety | duration of protocol

SECONDARY OUTCOMES:
pharmacokinetics | duration of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Benno G Roesch, MD, Principal Investigator — Advanced Biomedical Research, Inc.
Locations (1):
- Advanced Biomedical Research, Inc., Hackensack, New Jersey, United States